CLINICAL TRIAL: NCT05430438
Title: Effect of Low Versus Standard Dialysate Sodium on 48h Ambulatory BP in Patients With Intradialytic Hypertension
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aristotle University Of Thessaloniki (Other)
Responsible Party: Principal Investigator, Fotini Iatridi, Principal Investigator, PhD Candidate, Aristotle University Of Thessaloniki
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: ΔΔ4954
Record Dates: First submitted 2022-06-09; First posted 2022-06-24 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2023-09

CONDITIONS: Intradialytic Hypertension; End Stage Kidney Disease
Keywords: Intradialytic Hypertension; Dialysis; ESKD; Dialysate sodium
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Dialysis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): Patients will undergo dialysis (4 sessions) with low dialysate sodium (137 mEq/L) and after a 2-week washout period will undergo dialysis (4 sessions) with standard dialysis sodium (140 mEq/L).
  Interventions: Other: dialysis with low dialysate sodium concentration; Other: dialysis with standard dialysate sodium concentration
- Group B (Experimental): Patients will undergo dialysis (4 sessions) with standard dialysate sodium (140 mEq/L) and after a 2-week washout period will undergo dialysis (4 sessions) with low dialysis sodium (137 mEq/L).
  Interventions: Other: dialysis with low dialysate sodium concentration; Other: dialysis with standard dialysate sodium concentration

INTERVENTIONS:
Other: dialysis with low dialysate sodium concentration — Patients will undergo 4 dialysis sessions with a dialysate sodium concentration of 137 mEq/L. The modification of dialysate sodium concentration will be monitored through alteration of sodium conductivity
Other: dialysis with standard dialysate sodium concentration — Patients will undergo 4 dialysis sessions with a dialysate sodium concentration of 140 mEq/L. The modification of dialysate sodium concentration will be monitored through alteration of sodium conductivity

SUMMARY:
Intradialytic hypertension (IDH) is a well-recognized and established complication of hemodialysis that affects an estimated 10-15% of the dialysis population and is associated with an increased risk for cardiovascular adverse events and mortality. The major pathogenic mechanisms include volume and sodium overload, endothelial dysfunction and enhanced vasoconstriction potentially through the renin-angiotensin-aldosterone system (RAAS) and sympathetic nervous system (SNS) activation. Preliminary uncontrolled studies have demonstrated that in order to achieve proper control of blood pressure (BP) in patients with IDH, volume control with achievement of dry weight, as well as the minimization of sodium load through alteration of dialysate sodium may improve BP. To this day, 3 studies have attempted to evaluate the effect of low dialysate sodium on BP levels in patients with IDH; one study that included 16 patients, compared the effect of low (5 milliequivalent/litre (mEq/L) lower than serum sodium) versus high (5 mEq/L higher than serum sodium) dialysate sodium concentration on BP levels only during the dialysis session; another study examined the effect of low (136 mEq/L) compared to standard (140 mEq/L) sodium dialysate, again, only on peridialytic and intradialytic BP; and only one randomized cross-over study used 24h ABPM to assess the effect of individualized isonatremic vs hyponatremic vs standard dialysate sodium. Hence, the aim of this study is to examine the effect of low (137mEq/L) vs standard (140mEq/L) dialysate sodium on 48h ambulatory blood pressure monitoring (ABPM) in patients with IDH, using appropriate design of randomized crossover study. In addition this is the first study examining the effect of low dialysate sodium on ambulatory central BP, arterial stiffness indices and BP variability in patients with IDH.

DETAILED DESCRIPTION:
This is an interventional randomized crossover study performed in the Department of Nephrology, Hippokration Hospital, Thessaloniki, Greece. For the purposes of this study, adult patients (>18 years) with end stage kidney disease (ESKD) being treated with hemodialysis (HD) (on standard thrice-weekly HD treatment) for at least 3 months with intradialytic hypertension, fulfilling the inclusion/exclusion criteria were invited to participate. All included patients signed a written informed consent form. The study protocol was approved by the Ethics Committee of the School of Medicine, Aristotle University of Thessaloniki. All procedures and evaluations are performed according to the Declaration of Helsinki 2013 Amendment.

Patients will be assessed for eligibility during the selection process (records of peridialytic BP measurements of the previous 2-week period will be assessed). Patients will be instructed to arrive to the Dialysis unit 30 min to 1 hour prior to their scheduled dialysis session, on 3 different dialysis days. Baseline evaluation of participants includes the recording of demographics and anthropometric characteristics, medical history, comorbidities, concomitant medications and dialysis-related parameters, as well as physical examination and venous blood sampling for routine laboratory tests. At baseline evaluation patients' hydration status will be assessed with lung ultrasound, while peridialytic BP and BP over the intradialytic period will be assessed with the Mobil-O-Graph device (IEM, Stolberg, Germany). The study includes two treatment periods (low vs standard dialysate sodium) with washout period of 2 weeks between them. Patients will be randomized to 2 groups, which will receive the intervention in the opposite order. Block randomisation will be used to determine treatment order based on a computer-generated randomization list. The first group (A) will undergo dialysis with low dialysate sodium (137 mEq/L) for 4 sessions starting from a mid-week session (i.e Wednesday or Thursday). Immediately before the beginning of the 4th session patients will be assessed with lung ultrasound and the 48h ambulatory BP monitoring will start using the Mobil-O-Graph device. After a 2-week washout period this group (A) will undergo dialysis with standard dialysate sodium (140 mEq/L) for 4 sessions and at the start of the 4th session, again, patients will be assessed with lung ultrasound and the 48h ABPM will begin. The second group will undergo dialysis first with standard dialysate sodium (140 mEq/L) for 4 sessions and then, after the 2-week washout period, with low dialysate sodium (137 mEq/L) for 4 sessions, with similar evaluations at the end of each intervention. Patients will not be aware of the order in which they will receive the 2 different dialysate sodium concentrations.

ELIGIBILITY:
Inclusion Criteria:

* Adult ESKD individuals treated with a standard thrice weekly hemodialysis schedule for at least 3 months
* Patients with intradialytic hypertension, defined as SBP rise ≥10 mmHg from pre- to post-dialysis in at least 4 out of 6 consecutive sessions
* Patients that are considered clinically euvolemic
* Ability to provide informed written consent

Exclusion Criteria:

* Post-dialysis SBP <130 mmHg in at least 4 out of 6 consecutive sessions during the 2-week selection period, prior to study entry
* Previous non-functional arteriovenous fistula in the contralateral brachial arm area of the one used for vascular access that could interfere with proper ambulatory BP recording
* Patients with contraindications to receive the intervention (low dialysate sodium), i.e patients with frequent intradialytic hypotension episodes requiring intervention with fluid administration
* Pre-dialysis serum sodium <130 or >142 mEq/L at recruitment
* Modification of dry weight or antihypertensive treatment during one month before study initiation
* History of seizures or disequilibrium syndrome
* Hospitalization for any cause during one month before study initiation
* History of malignancy or any other condition with poor prognosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2023-07-24 (Actual); Study Completion 2023-07-24 (Actual)

PRIMARY OUTCOMES:
The difference in 48h ambulatory systolic blood pressure (SBP) between low and standard dialysate sodium in patients with intradialytic hypertension | At the 4th dialysis session and the following interdialytic interval of each intervention (end of weeks 2 and 5)

SECONDARY OUTCOMES:
The difference in 48h ambulatory diastolic blood pressure (DBP) between low and standard dialysate sodium in patients with intradialytic hypertension | At the 4th dialysis session and the following interdialytic interval of each intervention (end of weeks 2 and 5)
The difference in intradialytic SBP/DBP between low and standard dialysate sodium in patients with intradialytic hypertension | At the 4th dialysis session of each intervention (end of weeks 2 and 5)
The difference in pre-dialysis SBP/DBP between low and standard dialysate sodium in patients with intradialytic hypertension | At the 4th dialysis session of each intervention (end of weeks 2 and 5)
The difference in post-dialysis SBP/DBP between low and standard dialysate sodium in patients with intradialytic hypertension | At the 4th dialysis session of each intervention (end of weeks 2 and 5)
The difference in ambulatory aortic SBP/DBP between low and standard dialysate sodium in patients with intradialytic hypertension | At the 4th dialysis session and the following interdialytic interval of each intervention (end of weeks 2 and 5)
The difference in ambulatory Augmentation index (AIx) between low and standard dialysate sodium in patients with intradialytic hypertension | At the 4th dialysis session and the following interdialytic interval of each intervention (end of weeks 2 and 5)
The difference in ambulatory Augmentation index corrected for heart rate (AIx75) between low and standard dialysate sodium in patients with intradialytic hypertension | At the 4th dialysis session and the following interdialytic interval of each intervention (end of weeks 2 and 5)
The difference in ambulatory Augmentation pressure (AP) between low and standard dialysate sodium in patients with intradialytic hypertension | At the 4th dialysis session and the following interdialytic interval of each intervention (end of weeks 2 and 5)
The difference in ambulatory arterial stiffness between low and standard dialysate sodium in patients with intradialytic hypertension | At the 4th dialysis session and the following interdialytic interval of each intervention (end of weeks 2 and 5)
  Ambulatory arterial stiffness will be assessed by ambulatory pulse wave velocity (PWV), as recorded with the Mobil-O-Graph device
The difference in 48h ambulatory brachial SBP/DBP standard deviation (SD) between low and standard dialysate sodium in patients with intradialytic hypertension | At the 4th dialysis session and the following interdialytic interval of each intervention (end of weeks 2 and 5)
  This blood pressure variability (BPV) parameter of SBP/DBP will be calculated based on the ABPM recordings obtained with the Mobil-O-Graph device
The difference in 48h ambulatory brachial SBP/DBP weighted SD (wSD) between low and standard dialysate sodium in patients with intradialytic hypertension | At the 4th dialysis session and the following interdialytic interval of each intervention (end of weeks 2 and 5)
  This blood pressure variability (BPV) parameter of SBP/DBP will be calculated based on the ABPM recordings obtained with the Mobil-O-Graph device
The difference in 48h ambulatory brachial SBP/DBP coefficient of variation (CV) between low and standard dialysate sodium in patients with intradialytic hypertension | At the 4th dialysis session and the following interdialytic interval of each intervention (end of weeks 2 and 5)
  This blood pressure variability (BPV) parameter of SBP/DBP will be calculated based on the ABPM recordings obtained with the Mobil-O-Graph device
The difference in 48h ambulatory brachial SBP/DBP average real variability (ARV) between low and standard dialysate sodium in patients with intradialytic hypertension | At the 4th dialysis session and the following interdialytic interval of each intervention (end of weeks 2 and 5)
  This blood pressure variability (BPV) parameter of SBP/DBP will be calculated based on the ABPM recordings obtained with the Mobil-O-Graph device
The difference in pre-dialysis body weight between low and standard dialysate sodium in patients with intradialytic hypertension | At the 4th dialysis session of each intervention (end of weeks 2 and 5)
The difference in interdialytic weight gain (IDWG) between low and standard dialysate sodium in patients with intradialytic hypertension | At the 4th dialysis session of each intervention (end of weeks 2 and 5)
The difference in hydration status (b-lines) assessed by lung ultrasound between low and standard dialysate sodium in patients with intradialytic hypertension | At the 4th dialysis session of each intervention (end of weeks 2 and 5)
The difference (delta) between baseline and end-of-treatment values of each intervention for intradialytic SBP/DBP. | At baseline and at the 4th dialysis session of each intervention (baseline and end of weeks 2 and 5)
The difference (delta) between baseline and end-of-treatment values of each intervention for pre-dialysis SBP/DBP. | At baseline and at the 4th dialysis session of each intervention (baseline and end of weeks 2 and 5)
The difference (delta) between baseline and end-of-treatment values of each intervention for post-dialysis SBP/DBP. | At baseline and at the 4th dialysis session of each intervention (baseline and end of weeks 2 and 5)
The difference (delta) between baseline and end-of-treatment values of each intervention for pre-dialysis body weight. | At baseline and at the 4th dialysis session of each intervention (baseline and end of weeks 2 and 5)
The difference (delta) between baseline and end-of-treatment values of each intervention for IDWG. | At baseline and at the 4th dialysis session of each intervention (baseline and end of weeks 2 and 5)
The difference (delta) between baseline and end-of-treatment values of each intervention for hydration status (b-lines). | At baseline and at the 4th dialysis session of each intervention (baseline and end of weeks 2 and 5)
The difference between low and standard dialysate sodium in the delta for intradialytic SBP/DBP. | At baseline and at the 4th dialysis session of each intervention (baseline and end of weeks 2 and 5)
The difference between low and standard dialysate sodium in the delta for pre-dialysis SBP/DBP. | At baseline and at the 4th dialysis session of each intervention (baseline and end of weeks 2 and 5)
The difference between low and standard dialysate sodium in the delta for post-dialysis SBP/DBP. | At baseline and at the 4th dialysis session of each intervention (baseline and end of weeks 2 and 5)
The difference between low and standard dialysate sodium in the delta for pre-dialysis body weight. | At baseline and at the 4th dialysis session of each intervention (baseline and end of weeks 2 and 5)
The difference between low and standard dialysate sodium in the delta for IDWG. | At baseline and at the 4th dialysis session of each intervention (baseline and end of weeks 2 and 5)
The difference between low and standard dialysate sodium in the delta for hydration status (b-lines). | At baseline and at the 4th dialysis session of each intervention (baseline and end of weeks 2 and 5)

CONTACTS AND LOCATIONS:
Overall Officials: Pantelis Sarafidis, Prof, Study Director — Aristotle University Of Thessaloniki
Locations (4):
- Greece (3):
  - Frontis Dialysis Center, Athens
  - Therapeutiki Dialysis Unit, Thessaloniki
  - Aristotle University of Thessaloniki, Thessaloniki
- UKC Maribor, Maribor, Slovenia

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Georgianos PI, Sarafidis PA, Zoccali C. Intradialysis Hypertension in End-Stage Renal Disease Patients: Clinical Epidemiology, Pathogenesis, and Treatment. Hypertension. 2015 Sep;66(3):456-63. doi: 10.1161/HYPERTENSIONAHA.115.05858. Epub 2015 Jul 6. No abstract available. PMID 26150436
- [Background] Inrig JK, Molina C, D'Silva K, Kim C, Van Buren P, Allen JD, Toto R. Effect of low versus high dialysate sodium concentration on blood pressure and endothelial-derived vasoregulators during hemodialysis: a randomized crossover study. Am J Kidney Dis. 2015 Mar;65(3):464-73. doi: 10.1053/j.ajkd.2014.10.021. Epub 2014 Dec 17. PMID 25530107
- [Background] Nair SV, Balasubramanian K, Ramasamy A, Thamizhselvam H, Gharia S, Periasamy S. Effect of low dialysate sodium in the management of intradialytic hypertension in maintenance hemodialysis patients: A single-center Indian experience. Hemodial Int. 2021 Jul;25(3):399-406. doi: 10.1111/hdi.12921. Epub 2021 Mar 18. PMID 33733579
- [Background] Bikos A, Angeloudi E, Memmos E, Loutradis C, Karpetas A, Ginikopoulou E, Panagoutsos S, Pasadakis P, Liakopoulos V, Papagianni A, Sarafidis P. A Comparative Study of Short-Term Blood Pressure Variability in Hemodialysis Patients with and without Intradialytic Hypertension. Am J Nephrol. 2018;48(4):295-305. doi: 10.1159/000493989. Epub 2018 Oct 22. PMID 30347395
- [Background] Agarwal R, Light RP. Intradialytic hypertension is a marker of volume excess. Nephrol Dial Transplant. 2010 Oct;25(10):3355-61. doi: 10.1093/ndt/gfq210. Epub 2010 Apr 16. PMID 20400448
- [Background] Robberechts T, Allamani M, Galloo X, Wissing KM, Van Der Niepen P. Individualized Isonatremic and Hyponatremic Dialysate Improves Blood Pressure in Patients with Intradialytic Hypertension: A Prospective Cross-Over Study with 24-h Ambulatory Blood Pressure Monitoring. Open Journal of Nephrology 2020; 10:144-157
- [Background] Bikos A, Loutradis C, Angeloudi E, Karpetas A, Raptis V, Kalaitzidis R, Panagoutsos S, Pasadakis P, Balaskas I, Liakopoulos V, Papagianni A, Sarafidis PA. The effects of nebivolol and irbesartan on postdialysis and ambulatory blood pressure in patients with intradialytic hypertension: a randomized cross-over study. J Hypertens. 2019 Feb;37(2):432-442. doi: 10.1097/HJH.0000000000001891. PMID 30063644
- [Derived] Marshall MR, Wang MY, Vandal AC, Dunlop JL. Low dialysate sodium levels for chronic haemodialysis. Cochrane Database Syst Rev. 2024 Nov 5;11(11):CD011204. doi: 10.1002/14651858.CD011204.pub3. PMID 39498822
- [Derived] Iatridi F, Malandris K, Ekart R, Xagas E, Karpetas A, Theodorakopoulou MP, Karagiannidis A, Georgiou A, Papagianni A, Sarafidis P. Low dialysate sodium and 48-h ambulatory blood pressure in patients with intradialytic hypertension: a randomized crossover study. Nephrol Dial Transplant. 2024 Oct 30;39(11):1900-1910. doi: 10.1093/ndt/gfae104. PMID 38710537